CLINICAL TRIAL: NCT03525925
Title: Pilot Study Testing the Effects of BTK Inhibitor Ibrutinib on Levels and Function of Myeloid Derived Suppressor Cells and Other Immune Subsets in Patients With Metastatic Solid Tumors
Brief Title: Ibrutinib and Nivolumab in Treating Participants With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Robert Wesolowski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18015; NCI-2018-00423 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, nivolumab) (Experimental): Participants receive ibrutinib PO daily for 15 days. After 7 days receiving ibrutinib, participants receive nivolumab IV over 60 minutes on days 1 and 15. Courses with nivolumab repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I trial studies how well ibrutinib and nivolumab work in treating participants with solid tumors that have spread to other places in the body. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving ibrutinib and nivolumab may work better in treating participants with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of the ibrutinib therapy on circulating levels of myeloid derived suppressor cells MDSC.

SECONDARY OBJECTIVES:

I. Assess safety of the study combination in study subjects.

EXPLORATORY OBJECTIVES:

I. Evaluate the effect of the ibrutinib/nivolumab therapy on circulating levels of MDSC.

II. Evaluate the effect of the ibrutinib and ibrutinib/nivolumab therapy on the immunosuppressive function of circulating MDSC by measuring their ability to inhibit T cell proliferation and natural killer cell mediated antibody dependent cell cytotoxicity.

III. Study the effect of ibrutinib and ibrutinib/nivolumab therapy on levels of circulating innate and adaptive immune cells such as natural killer cell and T lymphocyte subsets.

IV. Study circulating MDSC levels at the time of disease progression. V. Evaluate in a preliminary fashion the effect of the regimen on progression-free survival.

OUTLINE:

Participants receive ibrutinib orally (PO) daily for 15 days. After 7 days receiving ibrutinib, participants receive nivolumab intravenously (IV) over 60 minutes on days 1 and 15. Courses with nivolumab repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, participants are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven metastatic solid tumor and be eligible to receive nivolumab per standard of care
* Patients will be allowed to have any number of prior lines of therapy for metastatic cancer
* Patients with measurable and non-measurable disease are allowed to participate
* Absolute neutrophil count (ANC) ? 1.5 x 10^3/mm^3
* Hemoglobin (Hgb) ? 9 g/dL
* Platelet count ? 100 x10^3/mm^3
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ? 2.5 x upper limit of normal (ULN) or ? 5 x ULN in patients with liver metastases
* Prothrombin time ? 1.5 x ULN
* Total bilirubin ? 1.5 x ULN (unconjugated bilirubin of < 3 x ULN for patients with known Gilbert syndrome)
* Creatinine clearance of ? 50 ml/min by Cockcroft-Gault equation
* Corrected QT interval of < 480 msec (using either Bazett?s or Fridericia's formula)
* Life expectancy of > 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ? 2
* Sexually active women with child bearing potential must have a negative pregnancy test obtained within 14 days prior to initiating study treatment
* Sexually active women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after completion of study treatment administration; adequate contraception includes methods such as oral contraceptives, double barrier method (condom plus spermicide or diaphragm), or abstaining from sexual intercourse

Exclusion Criteria:

* History of prior therapy with ibrutinib or nivolumab
* Unable to swallow capsules or having disease that is significantly affecting gastrointestinal function and/or inhibiting small intestine absorption
* Diagnosis of congenital or acquired immunodeficiency with the exception of chemotherapy induced immune suppression
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids of greater than or equal to prednisone 10 mg/day or other immunosuppressive agents; patients with history of adequately treated Hashimoto?s thyroiditis will be eligible; patients requiring a short course of a high dose prednisone burst to treat asthma or common obstructive pulmonary disease will also be eligible 5 days following completion of the prednisone treatment
* Use of systemic steroids at a dose above 10 mg/day of prednisone or prednisone equivalent in cycle 1 of study therapy; systemic steroids must be discontinued at least 5 days prior to initiating study therapy; exception will be given to patients who develop immune related adverse events that necessitate use of steroids or other immune suppressive agents; following cycle 1 of study treatment, the use of systemic steroids will be allowed per discretion of the treating physician
* Active, non-infectious pneumonitis
* Ongoing or active infection requiring systemic therapy
* History of being positive for human immunodeficiency virus (HIV)
* History of hepatitis B or C
* History of receiving live vaccine within 30 days of planned start of study therapy
* Central nervous system (CNS) metastases or leptomeningeal carcinomatosis; patients with history of adequately treated brain metastases that are stable for > 2 weeks prior to the first dose of study regimen are eligible as long they no longer require steroids and have no seizures or worsening focal neurologic symptoms; anti-epileptic therapy will be allowed
* Patients who had prior systemic chemotherapy within 3 weeks (or < 5 half-lives ? whichever is longer)
* Prior radiation therapy within 2 weeks of study enrollment
* Prior investigational therapy within 4 weeks
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to the first dose of study drug; port placement will not be considered major or minor surgery
* Any inter-current, uncontrolled systemic illness or any medical or psychiatric condition that in the opinion of the investigator would make the study therapy unsafe to the patient
* Unable to understand and sign informed consent form
* Uncontrolled, active cardiovascular disease including, but not limited to: symptomatic congestive heart failure, any class 3 or 4 cardiac disease as defined by the New York Heart Association functional classification, unstable angina pectoris, cardiac arrhythmia
* Any medications or substances that are strong inhibitors or inducers of CYP 3A4 need to be discontinued prior to initiation the study therapy and for the duration of ibrutinib treatment; patients can resume these medications 3 days after completion of ibrutinib course
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as ibrutinib or nivolumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Circulating levels of myeloid derived suppressor cells | Up to 2 years
  Will be summarized using descriptive statistics (N, mean, standard deviation, median, minimum, and maximum) and/or frequency and percentages for medically relevant categories. Changes of the continuous variables will be estimated using mixed model for repeated measures with proper data transformation as needed, and two-way tables and Chi-Square test will be used to summarize the changes of the categorical data.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Will be presented using frequencies and percentages.
Progression free survival | Interval from study enrollment to first documented disease progression according to Response Evaluation Criteria in Solid Tumors 1.1 or death from any cause (whichever occurs first), assessed at 1 year
  One year progression free survival will be defined as proportion of patients who are free of disease progression or death (whichever occurs first) after 1 year of follow up. Progression free survival will be summarized using Kaplan and Meier methods, where patients who are event-free at the time of their last evaluation will be censored at that time point.

OTHER OUTCOMES:
Biomarker analysis | Up to 2 years
  Will assess the association between the clinical responses and biomarkers/immune cell populations of interest will be identified using conventional techniques. These analyses will be primarily exploratory and hypothesis-generating. Will study the biomarker association with clinical outcomes using descriptive statistics, graphical methods and statistical modeling where appropriate. T-tests (continuous variables), chi-square or Fisher?s Exact tests (categorical variables), logistic regression models or Cox proportional hazard models will be used to explore associations between biomarkers/immune cell populations and clinical responses, whichever is appropriate. Pre and post treatment biomarkers will be compared using either paired t-tests or non-parametric tests if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wesolowski, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarz E, Benner B, Wesolowski R, Quiroga D, Good L, Sun SH, Savardekar H, Li J, Jung KJ, Duggan MC, Lapurga G, Shaffer J, Scarberry L, Konda B, Verschraegen C, Kendra K, Shah M, Rupert R, Monk P, Shah HA, Noonan AM, Bixel K, Hays J, Wei L, Pan X, Behbehani G, Hu Y, Elemento O, Chung D, Xin G, Blaser BW, Carson WE 3rd. Inhibition of Bruton's tyrosine kinase with PD-1 blockade modulates T cell activation in solid tumors. JCI Insight. 2024 Nov 8;9(21):e169927. doi: 10.1172/jci.insight.169927. PMID 39513363
- See also: The Jamesline — http://cancer.osu.edu